CLINICAL TRIAL: NCT02784743
Title: Impact of Albendazole -Ivermectin Combination Treatment on Wuchereria Bancrofti Infection and Transmission in Mali
Brief Title: Impact of Albendazole -Ivermectin on Wuchereria Bancrofti in Mali
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre d'Appui à la lutte contre la Maladie (Other)
Collaborators: Malaria Research and Training Center, Bamako, Mali (Other); World Health Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMS/TDR ID# A00563
Record Dates: First submitted 2015-04-29; First posted 2016-05-27 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Lymphatic Filariasis
Keywords: Wuchereria bancrofti; Anopheles; Albendazole; Ivermectin; MDA
MeSH Terms: conditions — Elephantiasis, Filarial | interventions — Albendazole; Ivermectin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- albendazole and ivermectin (Experimental): Before and after design with all eligible volunteers receiving the study drugs. Administration of a yearly unique dose of albendazole 400mg and ivermectin 150ug/kg weight ( according to the height).
  Interventions: Drug: ''albendazole'' and ''ivermectin''

INTERVENTIONS:
Drug: ''albendazole'' and ''ivermectin'' — annual single dose administration of albendazole 400mg and ivermectin 150ug/kg of weight (according to the height)
  Other Names: Zentel and Mectizan

SUMMARY:
Lymphatic filariasis is a public health problem in Mali. The existing data are not up to date and most of them are more than 15 years old. To address this issue in April 2000, the investigators started studies to update the epidemiology of lymphatic filariasis. There is no ongoing lymphatic filariasis control program in 2000 in Mali in terms of preventive chemotherapy treatment or vector control.

To fill these gaps, this current study aims to assess the impact of albendazole-ivermectin combination treatment on Wuchereria bancrofti infection and transmission in 6 rural highly endemic villages of Mali.

DETAILED DESCRIPTION:
Lymphatic filariasis is a public health problem in Mali. The existing data are not up to date and most of them are more than 15 years old. To address this issue in April 2000, the investigators started studies to update the epidemiology of lymphatic filariasis. As a result, in two rural areas (Banambani and Sirakoro) located at about 25 km North-East Bamako, the parasite prevalence using ICT cards in August 2000 were 16% (n=150) and 15.0% (n=113) respectively in Banambani and Sirakoro. There is no ongoing lymphatic filariasis control program in 2000 in Mali in terms of preventive chemotherapy treatment or vector control.

To fill these gaps, this current study aims to assess the impact of albendazole-ivermectin combination treatment on Wuchereria bancrofti infection and transmission in 6 rural highly endemic villages of Mali.

The study will be conducted in three phases: the pre treatment assessment of lymphatic filariasis infection and transmission parameters, treatment phase with annual single dose of albendazole and ivermectin and the post treatment assessment of Anopheles gambiae s.l mosquitoes, the transmission parameters of the vectors in the community, human infection prevalence post treatment using Giemsa -stained thick smears and others test like the Immuno chromatographic test (ICT).

ELIGIBILITY:
Inclusion Criteria:

* resident of the 6 villages
* 5 years and above

Exclusion Criteria:

* pregnant women
* breastfeeding women

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1139 (Actual)
Dates: Start 2001-05; Primary Completion 2008-12 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
vector infection and infectivity rates | up to 7 months
  vectors are collected with human landing catch technique and the presence of Wb larvae stage s assessed using dissection method

SECONDARY OUTCOMES:
Post MDA adverses events related to the drug albendazo and ivermectin | up to 12 months
  after the administration of the drug the investigators assess the reaction to the treatment
impact of albendazole ivermectin treatment on microfilaremia | up to 12 months
  night thick smears on eligible volunteers 5 years and above

CONTACTS AND LOCATIONS:
Overall Officials: Sékou F Traoré, PhD, Principal Investigator — Malaria Research and Training Center, Mali

REFERENCES:
- [Background] Coulibaly YI, Dembele B, Diallo AA, Konate S, Dolo H, Coulibaly SY, Doumbia SS, Soumaoro L, Coulibaly ME, Bockarie MJ, Molyneux D, Nutman TB, Klion AD, Toure YT, Traore SF. The Impact of Six Annual Rounds of Mass Drug Administration on Wuchereria bancrofti Infections in Humans and in Mosquitoes in Mali. Am J Trop Med Hyg. 2015 Aug;93(2):356-60. doi: 10.4269/ajtmh.14-0516. Epub 2015 Jun 1. PMID 26033027
- [Result] Coulibaly YI, Dembele B, Diallo AA, Kristensen S, Konate S, Dolo H, Dicko I, Sangare MB, Keita F, Boatin BA, Traore AK, Nutman TB, Klion AD, Toure YT, Traore SF. Wuchereria bancrofti transmission pattern in southern Mali prior to and following the institution of mass drug administration. Parasit Vectors. 2013 Aug 28;6(1):247. doi: 10.1186/1756-3305-6-247. PMID 23981378
- See also: Abstract of Baseline and first mass drug adminstration data — http://www.ncbi.nlm.nih.gov/pubmed/23981378